CLINICAL TRIAL: NCT06815250
Title: Effectiveness of the Influenza and Tdap (tetanus, Diphtheria, Acellular Pertussis) Vaccination Educational and Learning Module (InTroDuce-Programme) in Improving Knowledge and Future Uptake of Vaccination Among Pregnant Mothers in Primary Care Clinics: a Randomised Control Trial Secondary IDs
Brief Title: Enhancing Maternal Vaccine Knowledge and Uptake: the InTroDuce-Programme Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Lau Hung Chiun, Medical Lecturer and Family Medicine Specialist, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: InTroDuce-Programme
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Vaccination Uptake; Knowledge; Tetanus, Diphtheria and Acellular Pertussis Vaccination; Influenza; Web Based Intervention; Vaccine Knowledge
Keywords: Influenza vaccination; Tdap vaccination; Educational module; Pregnant mothers; Vaccine knowledge; Vaccine uptake
MeSH Terms: conditions — Tetanus; Diphtheria; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: web-based educational video on Influenza and Tdap vaccine (InTroDuce-Programme)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Standard antenatal care
- Intervention (Experimental): Influenza and Tdap Vaccination Web-based Educational and Learning Module (InTroDuce-Programme)
  Interventions: Behavioral: Influenza and Tdap Vaccination Educational and Learning Module

INTERVENTIONS:
Behavioral: Influenza and Tdap Vaccination Educational and Learning Module — Influenza and Tdap learning and educational module delivered via website. The module will cover importance of vaccination for both pregnant women and infant, safety and efficacy of the influenza and TdaP vaccines, timing of vaccination, and addressing common concerns and misconceptions.
  Arms: Intervention

SUMMARY:
The goal of this InTroDuce-Programme interventional trial aims to test whether a web-based educational program can improve pregnant women's knowledge about Influenza and Tdap vaccinations and increase their intention to get vaccinated in the future. The main questions it aims to answer are:

Does the InTroDuce-Programme increase knowledge and future intention of pregnant mothers to get vaccinated against Influenza and Tdap? How does demographic factors, attitudes and barriers affect vaccination decisions among pregnant mothers?

Researchers will compare InTroDuce-Programme to standard care (routine antenatal care) to see if InTroDuce-Programme works to improve knowledge and future intention of pregnant mothers to be vaccinated against Influenza and Tdap. Participants will:

Receive the web-based educational module (InTroDuce-Programme), which covers the importance, safety, and effectiveness of vaccinations, as well as addressing common concerns.

Be followed up one month after the intervention. Answer questionnaires before and after the intervention to measure changes in vaccination knowledge and future intention to get vaccinated

DETAILED DESCRIPTION:
1.0 Background and Significance

Maternal vaccination is a crucial public health strategy to protect mothers and infants from infectious diseases like influenza and pertussis. Pregnant women face higher risks of complications due to physiological and immunological changes, with a fourfold increased likelihood of influenza-related hospitalization. Similarly, pertussis is particularly severe in infants under two months. In Malaysia, the Ministry of Health recommends influenza and Tdap vaccines during pregnancy, but uptake remains low due to safety concerns, limited provider recommendations, and access issues. Digital interventions, particularly video-based education, have shown promise in addressing vaccine hesitancy. To tackle these barriers, the InTroDuce-Programme, a comprehensive web-based educational module, has been developed to improve vaccination knowledge and uptake.

2.0 Objective

General objective: To evaluate the effectiveness of the InTroDuce-Programme in improving knowledge and future uptake of influenza and Tdap vaccination among pregnant mothers.

Specific objectives:

1. To determine the sociodemographic factors and clinical variables among study population.
2. To determine the prevalence of future vaccination uptake following the InTroDuce-Programme.
3. To evaluate the level of participants' attitudes and barriers towards future vaccination uptake before and after the InTroDuce-Programme.
4. To determine the effectiveness of the InTroDuce-Programme in improving knowledge and future uptake of influenza and Tdap vaccination among pregnant mothers.
5. To determine the factors associated with low future uptake of vaccine with socio-demographic factors (age, race, income, education) among pregnant mothers.

3.0 Methodology

3.1 Study Design

This randomised controlled trial (RCT) will be conducted in four primary care clinics in Hulu Langat district which are Klinik Kesihatan Kajang, Klinik Kesihatan Bangi, Klinik Kesihatan Batu 9 and Klinik Kesihatan Balakong. The study duration is 12 months, with recruitment over 6 months. A second follow-up will be conducted one month after providing the InTroDuce-Programme. Two clinics will be randomly assigned to administer the InTroDuce-Programme, while the other two will be provided with standard care, in order to minimise contamination.

Cluster definition based on urban and suburban classification Klinik Kesihatan Kajang and Klinik Kesihatan Bangi are classified as urban, while Klinik Kesihatan Batu 9 and Klinik Kesihatan Balakong are classified as suburban. These clinics were selected due to their geographic and demographic similarity, coupled with variability in socioeconomic, educational, cultural, and attitudinal factors. This selection ensures a balanced representation of diverse populations, enhancing the generalizability and applicability of the study findings. The approach is particularly valuable for comprehensively understanding the factors that influence vaccine knowledge and uptake among pregnant mothers.

Random Allocation of Clinics Random Assignment: One clinic from each category (urban and suburban) will be randomly assigned to either the intervention or control group using an online random number generator. This method ensures unbiased allocation and maintains the balance of geographic representation in both groups.

The rationale for Randomization is to minimise contamination. Randomizing at the clinic level (cluster randomization) rather than at the individual level will help reduce the risk of contamination, where participants in the same clinic may share information or influence each other's behaviour. By assigning entire clinics to either intervention or control, the study ensures that participants within each clinic receive consistent and isolated exposure to the educational materials or standard care.

3.2 Sample Size

The sample size is 351 participants, accounting for a 20% non-response rate. This is based on expected uptake rates of 55% in the intervention group and 36% in the control group.

3.3 Data Collection

A validated, adapted questionnaire will be used in this study to assess vaccine-related knowledge, attitudes, future uptake intentions, and factors influencing vaccination decisions.

3.4 Statistical Analysis

Primary Outcome: Knowledge improvement, analyzed via paired t-tests or Mann-Whitney U tests.

Secondary Outcomes: Logistic regression for factors associated with low uptake intentions.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 years and older
* Before or equal to 32 weeks of gestation as we need to follow-up the patients again at 36 weeks of gestation before delivery occurs.
* Able to understand and consent to participation in the study.

Exclusion Criteria:

* Pregnant women with severe anaphylactic or allergic reactions to previous dose of influenza or Tdap vaccination.
* Non-Malaysian

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 351 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge of Influenza and Tdap Vaccination | 1 month post-intervention
  knowledge score about the importance, safety, and benefits of vaccination (vaccine literacy) will be assessed through pre- and post-intervention questionnaire
Vaccination Future Uptake | 1 month post-intervention
  Intention of future vaccine uptake of the influenza and Tdap vaccines will be assessed using questionnaire

SECONDARY OUTCOMES:
Barriers to vaccination uptake | 1 month post-intervention
  Identification of barriers to vaccination uptake and socio-demographic factors influencing outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Hung Chiun Lau, Dr Fam Med, Principal Investigator — Universiti Putra Malaysia
Locations (4):
- Malaysia (4):
  - Klinik Kesihatan Bangi, Bandar Baru Bangi, Selangor
  - Klinik Kesihatan Batu 9, Cheras, Selangor
  - Klinik Kesihatan Balakong, Cheras, Selangor
  - Klinik Kesihatan Kajang, Kajang, Selangor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Leary ST, Narwaney KJ, Wagner NM, Kraus CR, Omer SB, Glanz JM. Efficacy of a Web-Based Intervention to Increase Uptake of Maternal Vaccines: An RCT. Am J Prev Med. 2019 Oct;57(4):e125-e133. doi: 10.1016/j.amepre.2019.05.018. Epub 2019 Aug 27. PMID 31471001
- [Background] Deverall EJ, Gilmore B, Illing S, Peiris-John R. Pertussis vaccination uptake in pregnancy: lessons to be learned from an integrated healthcare approach. N Z Med J. 2018 Apr 13;131(1473):42-47. PMID 29649195
- [Background] Dawood FS, Kittikraisak W, Patel A, Rentz Hunt D, Suntarattiwong P, Wesley MG, Thompson MG, Soto G, Mundhada S, Arriola CS, Azziz-Baumgartner E, Brummer T, Cabrera S, Chang HH, Deshmukh M, Ellison D, Florian R, Gonzales O, Kurhe K, Kaoiean S, Rawangban B, Lindstrom S, Llajaruna E, Mott JA, Saha S, Prakash A, Mohanty S, Sinthuwattanawibool C, Tinoco Y. Incidence of influenza during pregnancy and association with pregnancy and perinatal outcomes in three middle-income countries: a multisite prospective longitudinal cohort study. Lancet Infect Dis. 2021 Jan;21(1):97-106. doi: 10.1016/S1473-3099(20)30592-2. Epub 2020 Oct 29. PMID 33129424
- [Background] Hong EY, Kulkarni K, Gosavi A, Wong HC, Singh K, Kale AS. Assessment of knowledge and attitude towards influenza and pertussis vaccination in pregnancy and factors affecting vaccine uptake rates: a cross-sectional survey. Singapore Med J. 2023 Aug;64(8):513-516. doi: 10.11622/smedj.2021097. No abstract available. PMID 34544209
- [Background] Razai MS, Mansour R, Goldsmith L, Freeman S, Mason-Apps C, Ravindran P, Kooner P, Berendes S, Morris J, Majeed A, Ussher M, Hargreaves S, Oakeshott P. Interventions to increase vaccination against COVID-19, influenza and pertussis during pregnancy: a systematic review and meta-analysis. J Travel Med. 2023 Dec 28;30(8):taad138. doi: 10.1093/jtm/taad138. PMID 37934788
- [Background] Kilich E, Dada S, Francis MR, Tazare J, Chico RM, Paterson P, Larson HJ. Factors that influence vaccination decision-making among pregnant women: A systematic review and meta-analysis. PLoS One. 2020 Jul 9;15(7):e0234827. doi: 10.1371/journal.pone.0234827. eCollection 2020. PMID 32645112
- [Background] Racicot K, Mor G. Risks associated with viral infections during pregnancy. J Clin Invest. 2017 May 1;127(5):1591-1599. doi: 10.1172/JCI87490. Epub 2017 May 1. PMID 28459427
- [Background] Arora M, Lakshmi R. Vaccines - safety in pregnancy. Best Pract Res Clin Obstet Gynaecol. 2021 Oct;76:23-40. doi: 10.1016/j.bpobgyn.2021.02.002. Epub 2021 Feb 19. PMID 33773923
- [Background] Merdrignac L, Acosta L, Habington A, Garcia Cenoz M, Pandolfi E, Fabianova K, Jordan I, O'Sullivan N, Navasues A, Tozzi AE, Zavadilova J, Jane M, Cotter S, Pitillas NI, Rizzo C, Krizova P, Hanslik T, Munoz Almagro C, Pastore L, Bacci S, Moren A, Valenciano M; PERTINENT Group. Effectiveness of pertussis vaccination in pregnancy to prevent hospitalisation in infants aged <2 months and effectiveness of both primary vaccination and mother's vaccination in pregnancy in infants aged 2-11 months. Vaccine. 2022 Oct 19;40(44):6374-6382. doi: 10.1016/j.vaccine.2022.09.054. Epub 2022 Sep 29. PMID 36182617
- [Background] Razai MS, Mansour R, Ravindran P, Freeman S, Mason-Apps C, Morris J, Majeed A, Ussher M, Hargreaves S, Oakeshott P. Facilitators and barriers to vaccination uptake in pregnancy: A qualitative systematic review. PLoS One. 2024 Apr 19;19(4):e0298407. doi: 10.1371/journal.pone.0298407. eCollection 2024. PMID 38640190
- [Background] Razai MS, Chaudhry UAR, Doerholt K, Bauld L, Majeed A. Covid-19 vaccination hesitancy. BMJ. 2021 May 20;373:n1138. doi: 10.1136/bmj.n1138. No abstract available. PMID 34016653
- [Background] Parsons J, Griffiths SE, Thomas N, Atherton H. How effective are digital interventions in increasing flu vaccination among pregnant women? A systematic review and meta-analysis. J Public Health (Oxf). 2022 Dec 1;44(4):863-876. doi: 10.1093/pubmed/fdab220. PMID 34164686
- See also: Centers for Disease Control and Prevention (CDC). (2023). Vaccination During Pregnancy — https://www.cdc.gov/vaccines-pregnancy/about/index.html
- See also: PERINATAL CARE MANUAL 4th EDITION. Ministry of Health. 2022 — https://hq.moh.gov.my/bpkk/images/PERINATAL_CARE_MANUAL_4th_Edition_2020_11Mei2023.pdf